CLINICAL TRIAL: NCT04230421
Title: Effects of Smartphone-based Treatment for Bipolar Disorder - the Smart Bipolar RCT
Brief Title: Effects of Smartphone-based Treatment for Bipolar Disorder - the Smart Bipolar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Maria Faurholt-Jepsen, MD, DMSc (Unknown); The Mental Health Services in the Capital Region of Denmark (Unknown)
Responsible Party: Principal Investigator, Lars Vedel Kessing, Prof., Principal Investigator, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-19067259
Record Dates: First submitted 2020-01-03; First posted 2020-01-18 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monsenso with feedback (Experimental): Daily smartphone-based monitoring and treatment using the Monsenso system with a clinical feedback loop feedback.
  Interventions: Device: The Monsenso system with feedback
- Monsenso without feedback (Active Comparator): Daily smartphone-based monitoring and treatment using the Monsenso system WITHOUT a clinical feedback loop feedback.
  Interventions: Device: The Monsenso system without feedback
- Control (Active Comparator): CAG Bipolar treatment alone and daily mood monitoring using only the mood monitoring part of the Monsenso system.
  Interventions: Device: CAG Bipola and mood monitoring only

INTERVENTIONS:
Device: The Monsenso system with feedback — See description under intervention
  Arms: Monsenso with feedback
Device: The Monsenso system without feedback — See description under intervention
  Arms: Monsenso without feedback
Device: CAG Bipola and mood monitoring only — See description under intervention
  Arms: Control

SUMMARY:
The Smart Bipolar RCT is a pragmatic RCT aiming to investigate effects of smartphone-based add on treatment in large scale clinical practice (N= 200 patients).

DETAILED DESCRIPTION:
Bipolar disorder is a complex illness with a complex treatment that differs during manic, depressed, and remitted states, frequently leaving patients with decreased quality of life and impaired psychosocial function. IT solutions have during recent years emerged as a possible way to optimize treatment, but the effects of digital health interventions are rarely investigated scientifically in health care services.

This is an application from the entire Mental Health Services, Capital Region of Denmark including all psychiatric centers in the region. The Smart Bipolar randomized controlled trial is a pragmatic trial aiming to investigate the effects of smartphone-based add-on treatment in large-scale clinical practice (N= 200 patients). Findings from the study will have a great impact on future IT monitoring and treatment in bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* All patients in CAG Bipolar, i.e., with a main diagnosis of bipolar disorder in the five large centers, in the Mental Health Services, Capital Region of Denmark (Psychiatric Center Copenhagen, Psychiatric Center Hilleroed, Psychiatric Center Amager, Psychiatric Center Glostrup and Psychiatric Center Ballerup)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Daily self-reported mood instability via Monsenso | During the entire study period of 6 months per participant
  Mood measured daily via smartphones on a scale form -3 to +3.

SECONDARY OUTCOMES:
Risk of psychiatric hospitalization | During the entire study period of 6 months per participant
  Data on hospitalization according to data from the population-based Danish Psychiatric Central Research Register will be collected and analyzed with survival statistics. Assessed blinded for the intervention status.
Cumulated duration of psychiatric hospitalization | During the entire study period of 6 months per participant
  Data on hospitalization according to data from the population-based Danish Psychiatric Central Research Register will be collected and analyzed with survival statistics. Assessed blinded for the intervention status.
Quality of life according to WHO Quality of Life-BREF | Baseline and 6 months
  Scored between 0-100. Higher scores indicate higher quality of life. Patient evaluated
Patient-evaluated depressive symptoms according to the Major Depressive Inventory | Baseline and 6 months
  Higher scores indicate higher severity of depressive symptoms. Patient evaluated.
Patient-evaluated manic symptoms according to the Altman Self-rating Scale for Mania | Baseline and 6 months
  Higher scores indicate higher severity of manic symptoms. Patient evaluated.
Perceived stress according to Cohen's Perceived stress scale | Baseline and 6 months
  Patient evaluated. Scores between 0-40. Higher score indicate higher perceived stress.
Satisfaction with care according to scores on the Verona Satisfaction Scale-Affective Disorder | Baseline and 6 months
  Patient evaluated. Higher scores indicate higher satisfaction with treatment.
Adherence to the Danish national guidelines of medical treatment of bipolar disorder according to use of the three main maintenance mood stabilizers for bipolar disorder: lithium, lamotrigine or quetiapine and the use of antidepressants | During the entire study period of 6 months
  Adherence to medication will be an additional outcome measure in arms 1 and 2 of the RCT based on daily self-monitoring of medication via the Monsenso system.

OTHER OUTCOMES:
Patient-reported smartphone-based symptoms | During the entire study period of 6 months
  Patietns-reported smartphone-based symptoms such as stress, anxiety, activity, sleep, mixed mood, adherence to medication and adherence to patient-reported smartphone-based monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Center Copenhagen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faurholt-Jepsen M, Kyster NB, Dyreholt MS, Christensen EM, Bondo-Kozuch P, Lerche AS, Smidt B, Knorr U, Brondmark K, Cardoso AB, Mathiesen A, Sjaelland R, Norbak-Emig H, Sponsor LL, Mardosas D, Sarauw-Nielsen IP, Bukh JD, Heller TV, Frost M, Iversen N, Bardram JE, Busk J, Vinberg M, Kessing LV. The effect of smartphone-based monitoring and treatment including clinical feedback versus smartphone-based monitoring without clinical feedback in bipolar disorder: the SmartBipolar trial-a study protocol for a randomized controlled parallel-group trial. Trials. 2023 Sep 12;24(1):583. doi: 10.1186/s13063-023-07625-1. PMID 37700334